CLINICAL TRIAL: NCT01344837
Title: The Role of Synuclein-gamma (SNCG) in the Carcinogenesis of Uterine Papillary Serous Carcinoma
Brief Title: Biomarkers in Blood and Tissue Samples From Patients With Uterine Cancer
Status: Completed | Type: Observational
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Other Study IDs: GOG-8023; NCI-2011-02872 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000698458; GOG-8023 (Other: Gynecologic Oncology Group); GOG-8023 (Other: CTEP); R21CA135467 (NIH); U10CA027469 (NIH); U10CA037517 (NIH)
Record Dates: First submitted 2011-04-28; First posted 2011-04-29 (Estimated); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Endometrial Serous Adenocarcinoma; Stage I Uterine Corpus Cancer; Stage II Uterine Corpus Cancer; Stage III Uterine Corpus Cancer; Stage IV Uterine Corpus Cancer
MeSH Terms: interventions — Immunohistochemistry; Microarray Analysis; Transcriptome; Gene Expression Profiling; Blotting, Western

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Observational: Archived serum and tumor tissue samples are analyzed for synuclein-γ (SNCG) expression and other biomarker expression, including TP53 (p53), HER-2, folate receptor alpha (FOLR1), estrogen receptor (ER), progesterone receptor (PR), phosphatase and tensin homolog (PTEN), phosphorylated AKT (pAKT), pERK, and p16 by microarray analysis, IHC assays, and western blot. Results are then compared with patients' existing clinical, demographic, and pathology data, including history of breast cancer (metachronous) or breast cancer diagnosed at the same time as the endometrial cancer (synchronous).
  Interventions: Other: Diagnostic Laboratory Biomarker Analysis; Other: Immunohistochemistry Staining Method; Other: Medical Chart Review; Genetic: Microarray Analysis; Other: Study of Socioeconomic and Demographic Variables; Genetic: Western Blotting

INTERVENTIONS:
Other: Diagnostic Laboratory Biomarker Analysis — Correlative studies
Other: Immunohistochemistry Staining Method — Correlative studies
  Other Names: Cell/Tissue, Immunohistochemistry; IHC; Immunohistochemistry
Other: Medical Chart Review — Correlative studies
  Other Names: Chart Review
Genetic: Microarray Analysis — Correlative studies
  Other Names: gene expression profile; Gene Expression Profiling; Microarray Technology; Microarray-Based Analysis
Other: Study of Socioeconomic and Demographic Variables — Correlative studies
Genetic: Western Blotting — Correlative studies
  Other Names: Blotting, Western; WESTERN BLOT

SUMMARY:
This research study is studying biomarkers in blood and tissue samples from patients with uterine cancer. Studying samples of blood and tissue from patients with cancer in the laboratory may help doctors learn more about changes the occur in DNA and identify biomarkers related to cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine whether synuclein-γ (SNCG) expression in primary tumor is associated with overall survival (OS) in uterine papillary serous carcinoma (UPSC) patients.

SECONDARY OBJECTIVES:

I. Determine whether SNCG expression is associated with clinical covariates (age at diagnosis, race, surgical stage, depth of myometrial invasion, presence of lymph vascular space invasion, lymph node status, location of extrauterine disease, chemotherapy, and radiation therapy) in UPSC patients.

II. Determine whether SNCG expression is associated with other biomarker expression, including TP53 (p53), HER-2, folate receptor alpha (FOLR1), estrogen receptor (ER), progesterone receptor (PR), phosphatase and tensin homolog (PTEN), phosphorylated AKT (pAKT), pERK, and p16 in primary tumor tissue.

III. Determine whether SNCG expression is associated with progression-free survival (PFS).

IV. Determine whether SNCG expression is associated with synchronous or metachronous breast cancers.

EXPLORATORY OBJECTIVES:

I. Determine whether SNCG can be detected in sera from UPSC patients. II. Determine whether serum SNCG in UPSC patients differs from that in normal healthy control women and women with endometrioid endometrial cancer.

III. Determine whether serum SNCG in UPSC patients is associated with overall survival (OS), clinical covariates (listed above), tumor expression of biomarkers (listed above), PFS, and synchronous or metachronous breast cancers.

IV. Develop prediction models with a panel of biomarkers and clinical prognostic factors for OS, PFS, and synchronous or metachronous breast cancers in UPSC patients.

OUTLINE:

Archived serum and tumor tissue samples are analyzed for synuclein-γ (SNCG) expression and other biomarker expression, including TP53 (p53), HER-2, folate receptor alpha (FOLR1), estrogen receptor (ER), progesterone receptor (PR), phosphatase and tensin homolog (PTEN), phosphorylated AKT (pAKT), pERK, and p16 by microarray analysis, IHC assays, and western blot. Results are then compared with patients' existing clinical, demographic, and pathology data, including history of breast cancer (metachronous) or breast cancer diagnosed at the same time as the endometrial cancer (synchronous).

ELIGIBILITY:
Inclusion Criteria:

* Women with uterine papillary serous carcinoma (UPSC) who were eligible for GOG-0210 protocol, a molecular staging study in endometrial cancer, or GOG-0136, a general specimen banking study for gynecologic cancer, have consented to future research, have histologically-confirmed UPSC of any stage, and have satisfactory formalin-fixed and paraffin-embedded primary tumor with or without a satisfactory pre-operative serum specimen available for testing
* Women with endometrioid endometrial cancer who were eligible for GOG-0210 or GOG-0136, have consented to future research, have histologically-confirmed endometrioid endometrial carcinoma with a similar stage, age and race/ethnicity distribution as the UPSC patients, have satisfactory formalin-fixed and paraffin-embedded primary tumor and/or pre-operative serum specimen available for testing
* Normal healthy control women who participated in the Biopathology protocol for banking sera from normal healthy control women, have consented to future research, do not have a cancer or a history of cancer and have a similar age and race/ethnicity distribution as the UPSC patients and have satisfactory serum available for testing

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with uterine cancer
Sampling Method: Non-Probability Sample
Enrollment: 360 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Overall survival | From time of entry onto GOG-0210, assessed up to 2 years
  Kaplan-Meier survival curves for the overall survival (OS) endpoint will be generated separately for the three SNCG expression groups and globally compared using a log-rank test.

SECONDARY OUTCOMES:
Presence of synchronous or metachronous breast cancer | Up to 2 years
  Cox proportional hazards models with dummy variable coding of the SNCG expression groups will be used to estimate hazard ratios, with tests of interaction with time and log-log plots used to evaluate the proportional hazards assumption. Sensitivity of the estimated hazard ratios to adjustment for other variables will be explored in the analyses for the Secondary Objectives.
Progression-free survival | From time of entry onto GOG-0210 to time of progression, assessed up to 2 years
  Median survival times and 95% confidence intervals will be estimated from the Kaplan-Meier curves using Greenwood's formula for variance estimation.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Buttin, Principal Investigator — Gynecologic Oncology Group
Locations (1):
- Gynecologic Oncology Group, Philadelphia, Pennsylvania, United States